CLINICAL TRIAL: NCT05044845
Title: Needs Assessment of Knowledge, Beliefs, and Attitudes of Patients With Hemophilia B About Gene Therapy Globally
Brief Title: Needs Assessment of Knowledge, Beliefs, and Attitudes of Patients With Hemophilia B About Gene Therapy
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BINFORMED
Record Dates: First submitted 2021-09-09; First posted 2021-09-16 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Gene Therapy; Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hemophilia B patients: Patients ≥12 years of age with a diagnosis of moderate (FIX ≥1% and ≤2%) or severe (<1%) hemophilia B
  Interventions: Behavioral: Interview
- Parents or Caregivers: Parents or caregivers to patients with hemophilia 12-17 years of age
  Interventions: Behavioral: Interview
- Healthcare Workers: Doctors, nurses, social workers, pharmacists and educators who participate in the care of hemophilia B patients
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Semi structured interview will be conducted virtually using an online video-conferencing platform, phone or in person.
  Other Names: Questions

SUMMARY:
Gene therapy is a paradigm-shifting treatment for hemophilia B patients, particularly in resource-limited countries where factor availability remains low. Transparent and culturally sensitive communication around gene therapy is vital to the success of a high-quality consenting process. Current literature on knowledge, beliefs and attitudes about gene therapy in resource-limited countries is inadequate. In addition, few educational resources to explain basic gene therapy concepts exist in languages other than English. This study aims to address these gaps in knowledge and aid for the development of educational resources to assist the informed consent processes for gene therapy in resource-limited countries.

Primary Objective:

To assess baseline knowledge, beliefs, and attitudes about gene therapy held by hemophilia B patients globally

Secondary Objectives:

1. To explore healthcare workers' (i.e., physicians, nurses, social workers, educators/academic coordinators) perspectives regarding the education needs of hemophilia B patients globally
2. To explore healthcare workers beliefs and attitudes about gene therapy
3. To identify preferences of patients with hemophilia B and their healthcare workers on how/by what method or pathway educational content should be provided.

DETAILED DESCRIPTION:
This prospective cohort study will use qualitative methods, specifically semi structured interviews to evaluate knowledge, beliefs, and attitude about gene therapy in patients 12 years and older with a diagnosis of moderate and severe hemophilia B (≤2% FIX activity only), caregivers/parents and healthcare workers who care for them at St. Jude and other global countries. Participants will be interviewed virtually using an online video-conferencing platform, phone or in person.

Interviews will be performed by experienced qualitative interviewers in the official language of each participating site. Interviews will last approximately 45-60 minutes and will be performed only once. All interviews will be audio recorded and obtained information will be analyzed using semantic content analysis to identify common themes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥12 years of age
* Diagnosis of moderate (FIX ≥1% and ≤2%) or severe (<1%) hemophilia B
* Parents or caregivers to patients with hemophilia 12-17 years of age

Inclusion Criteria - Healthcare worker:

- Doctors, nurses, social workers, pharmacists and educators who participate in the care of hemophilia B patients

Exclusion Criteria:

* Diagnosis of Hemophilia A
* Diagnosis of other non-Hemophilia B bleeding disorders

Exclusion Criteria - Healthcare worker:

* Health care workers who do not participate in the care of hemophilia B patients
* Healthcare worker who is conducting the interviews

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Use of semi-structured interviews to qualitatively describe their attitudes, beliefs, and knowledge of gene therapy in hemophilia B | Day 1, or at a future visit (up to approximately 1 year)
  Semi-structured interviews will be performed in patients with hemophilia B, their caregivers and healthcare workers to qualitatively describe their attitudes, beliefs, and knowledge of gene therapy in hemophilia B including concerns, expectations, and best way to receive information about gene therapy. Interviews will be audio recorded, transcribed verbatim and analyzed using semantic content analysis to identify common themes.

CONTACTS AND LOCATIONS:
Overall Officials: Nidhi Bhatt, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (6):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States
- Civil Service Hospital, Kathmandu, Nepal
- Hospital Dos De Mayo, Lima, Peru
- National Hospital of Sri Lanka, Colombo, Sri Lanka
- Ramathibodi Hospital, Bangkok, Thailand
- National Institute of Hematology and Blood Transfusion, Hanoi, Vietnam

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols